CLINICAL TRIAL: NCT05117840
Title: Screening for High Frequency Malignant Disease
Acronym: SHIELD
Status: Active, not recruiting | Type: Observational
Sponsor: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 02-MX-002
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
Keywords: Screening; Non-invasive diagnostics
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draws will be taken and analyzed for all participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Cancer Screening Cohort: Individuals at high-risk of lung cancer undergoing standard of care screening as per USPSTF guidelines. All subjects will undergo low-dose CT scanning as per guidelines and an investigational blood-draw will be taken from all enrolled subjects.
  Interventions: Device: Low-dose CT scan

INTERVENTIONS:
Device: Low-dose CT scan — Standard of care screening for individuals at high-risk of lung cancer

SUMMARY:
The SHIELD (Screening for High Frequency Malignant Disease) study is a prospective, observational, multi-site basket design trial without randomization. The primary objective of the study is to evaluate the sensitivity and specificity of a blood-based GuardantLUNAR-2 test to detect high frequency cancer in screen-relevant populations.

DETAILED DESCRIPTION:
The SHIELD (Screening for High Frequency Malignant Disease) study is a prospective, observational, multi-site basket design trial without randomization. The primary objective of the study is to evaluate the sensitivity and specificity of a blood-based GuardantLUNAR-2 test to detect high frequency cancer in screen-relevant populations.

The SHIELD study will recruit patients in separate cancer-risk cohorts with specified pathways for cancer screening. Patients eligible for high frequency cancer screening will be screened for study eligibility per each cohort's criteria (see appendixes). Within each cohort, individuals eligible for the study will be consented for the investigational blood draw and applicable questionnaires within 90 days of standard of care screening method and prior to any invasive procedure for cancer diagnosis and/or treatment (T0). Subjects will have at least 2 follow-up visits at 1 year and 2 years (T1 and T2) since the index blood draw during the study. Additional follow-up is defined per each cohort. Updated medical data, repeat investigational blood draw and study questionnaires will be collected at follow-up intervals per each cohort's study procedure.

The first cohort to be recruited will be designated as cohort A for lung cancer screening (appendix 1). Additional baskets with other cancer-risk cohorts of interest will be considered and added as the study expands. Additional appendixes will be designed for these cohorts at that time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 50-80 years at time of consent
* Increased risk of lung cancer defined by: at least 20 pack-year smoking history and currently smoke or have quit within the past 15 years
* Undergoing or intended to undergo low dose CT scan of the chest for lung cancer screening
* Willing to consent to the investigational blood draw during index LDCT screening visit and before any invasive procedures or treatment for lung cancer diagnosis
* Willing to consent to a 1-year and additional follow-up per protocol

Exclusion Criteria:

1. Subject has quit smoking for 15 or more years
2. Subject has less than 20 pack-year smoking history
3. Subject has a health problem that substantially limits life expectancy and/or the ability or willingness to have curative lung surgery
4. Subject undergoing low-dose CT scan of the chest for investigation of symptoms suspicious for lung cancer
5. Preexisting or history of lung cancer
6. Previously diagnosed high-risk lung lesion
7. History of any malignancy (subjects who have undergone surgical removal of skin squamous cell cancer may be enrolled provided the procedure was completed at least 12 months prior to the date of provision of informed consent for the study)
8. Currently taking any anti-neoplastic or disease-modifying anti-rheumatic drugs
9. Currently receiving treatment for pneumonia
10. Any major physical trauma (e.g., disruption of tissue, surgery, organ transplant, blood product transfusion) within the 30 days leading up to the provision of informed consent
11. Known medical condition which, in the opinion of the investigator, should preclude enrollment into the study
12. Participation in a clinical research study in which an experimental medication and/or medical procedure has been administered or may be administered within the 30 days leading up to providing informed consent or may be administered through the time of subject screening

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The SHIELD study will recruit patients in separate cancer-risk cohorts with specified pathways for cancer screening. Patients eligible for high frequency cancer screening will be screened for study eligibility per each cohort's criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Performance characteristics of Guardant LUNAR-2 test | 36 months
  Sensitivity, specificity, NPV, PPV

SECONDARY OUTCOMES:
Screen detected cancer rate | 36 months
  To estimate the number of screen detected cancers, early-stage and late-stage screen detected cancers per 1000 screened subjects

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Oakley, Study Director — Guardant Health, Inc.
Locations (140):
- United States (122):
  - University of Alabama Birmingham Lung Health Center, Birmingham, Alabama
  - Highlands Oncology Group PA, Fayetteville, Arkansas
  - Pacific Cancer Medical Center, Anaheim, California
  - Providence St. Joseph Hospital Eureka Cancer Program, Eureka, California
  - SoCal Clinical Research, Fountain Valley, California
  - Advanced Investigative Medicine, Hawthorne, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Medical Research Associates Inc., Northridge, California
  - Providence Medical Foundation, Santa Rosa, California
  - Starling Physicians, New Britain, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Central Florida Pulmonary Group, P.A., Altamonte Springs, Florida
  - Pulmonary, Critical Care & Sleep Disorders Institute of South Florida, Atlantis, Florida
  - CTMD Research, Coconut Creek, Florida
  - Life Arc Research Centers, Coral Gables, Florida
  - Pulmonary Physicians of South Florida, LLC, Coral Springs, Florida
  - SIMED Health, LLC, Gainesville, Florida
  - National Research Institute, Hialeah, Florida
  - 3Sync Research, Hialeah, Florida
  - Zenith Clinical Research, Hollywood, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - 3Sync Research, Lake Worth, Florida
  - Adtremed INC, Lutz, Florida
  - Las Mias Research and Medical Center, Miami, Florida
  - Monzon Clinical Trials, Miami, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Miami Pulmonary Specialists, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Charisma Medical and Research Center, Miami Lakes, Florida
  - Adult Medicine of Lake County, Mt. Dora, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - CTMD Research, Palm Springs, Florida
  - Coastal Pulmonary and Critical Care, P.L.C., St. Petersburg, Florida
  - Adtremed Research Clinic, Tampa, Florida
  - VICIS Clinical Research, Tampa, Florida
  - Midtown OB/GYN North, Columbus, Georgia
  - Pulmonary and Sleep Specialists of Northeast Georgia, PC, Dacula, Georgia
  - DC Research Works, Marietta, Georgia
  - Randomize Now, LLC, Peachtree City, Georgia
  - Pulmonary and Sleep Specialists of Northeast Georgia, PC, Winder, Georgia
  - Christie Clinic, Champaign, Illinois
  - Eagle Clinical Research, Chicago, Illinois
  - Hutchinson Clinic - North Waldron, Hutchinson, Kansas
  - MedCorps Asthma and Pulmonary Specialists, Maysville, Kentucky
  - Family Medicine Physicians, Hammond, Louisiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - HealthPartners Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Family Medical Clinic of North Mississippi, Southaven, Mississippi
  - Branson Pulmonology and Sleep Medicine, Branson, Missouri
  - Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - Great Plains Health, North Platte, Nebraska
  - Ocean Pulmonary Associates, Brick, New Jersey
  - Ocean University Medical Center, Brick, New Jersey
  - RespaCare, Bridgewater, New Jersey
  - MedCorps Asthma and Pulmonary Specialists, Cape May Court House, New Jersey
  - Pulmonary & Sleep Disorders of New Jersey, East Brunswick, New Jersey
  - JFK University Medical Center, Edison, New Jersey
  - Pulmonary Internists, Edison, New Jersey
  - Pulmonary Specialists of North Jersey, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - MedCorps Asthma and Pulmonary Specialists, Linwood, New Jersey
  - Pulmonary & Sleep Disorders of New Jersey, Monroe, New Jersey
  - John Theurer Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Pulmonary Specialists of North Jersey, North Bergen, New Jersey
  - Respiratory and Sleep Specialists, LLC, Princeton, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - North Jersey Pulmonary Associates, Ridgewood, New Jersey
  - MedCorps Asthma and Pulmonary Specialists, Sewell, New Jersey
  - Ocean Pulmonary Associates, Toms River, New Jersey
  - Long Island Pulmonary and Sleep Medicine Associates, Hempstead, New York
  - Long Island Pulmonary and Sleep Medicine Associates, Rockville Centre, New York
  - Great Lakes Medical Research, Westfield, New York
  - CTMD Research, Asheville, Asheville, North Carolina
  - MacGregor Family Physicians, P.A., Cary, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Pulmonology Associates Inc., Broomall, Pennsylvania
  - Advocare Pulmonary And Sleep Specialists, Exton, Pennsylvania
  - Advocare Pulmonary And Sleep Specialists, Lansdale, Pennsylvania
  - Pulmonology Associates Inc., Paoli, Pennsylvania
  - Advocare Pulmonary And Sleep Specialists, West Chester, Pennsylvania
  - Pulmonology Associates Inc.Pulmonology Associates Inc. (Suite 108), Wynnewood, Pennsylvania
  - Pulmonology Associates Inc., Wynnewood, Pennsylvania
  - Berks Schuylkill Respiratory Specialists, Ltd., Wyomissing, Pennsylvania
  - Vista Clinical Research, Columbia, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Midsouth Independent Group, Memphis, Tennessee
  - MidSouth Independent Group, Memphis, Tennessee
  - Mid-South Pulmonary & Sleep Specialists PC, Memphis, Tennessee
  - Peabody Internal Medicine Inc., Millington, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Premier Family Physicians, Austin, Texas
  - ARC Clinical Research at William Cannon, Austin, Texas
  - Pulmonary Critical Care & Sleep Associates, P.A., Conroe, Texas
  - Horizon Clinical Research Group, Cypress, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - El Paso Pulmonary Associates, El Paso, Texas
  - Allure Heath at Mt. Olympus Medical Research, Friendswood, Texas
  - Best Cancer Care & Hematology - Biopharma Informatic, Houston, Texas
  - Huntsville Research Institute, LLC, Huntsville, Texas
  - Vytalus Medical Group, Kingwood, Texas
  - Covenant Health System/Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Wellness Clinical Research, McKinney, Texas
  - PRX Research, Mesquite, Texas
  - Oak Cliff Research, Richardson, Texas
  - Sugar Lakes Family Practice, PA, Sugar Land, Texas
  - Tidewater Physicians Multispecialty Group, P.C., Williamsburg, Virginia
  - Western Washington Medical Group, Inc, Everett, Washington
  - The Vancouver Clinic, Vancouver, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - Mayo Clinic Health System Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic La Crosse, La Crosse, Wisconsin
- France (12):
  - Centre Hospitalier d'Abbeville, Abbeville
  - CHU Amiens Picardie - Centre de Recherche Clinique, Amiens
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - Hopital Europeen, Marseille
  - Hopital Pasteur CHU de Nice de Pneumologie, Nice
  - Hõpital Lyon Sud, Pierre-Bénite
  - Saint-Quentin Hospital Center, Saint-Quentin
  - Hôpitaux du Léman, Thonon-les-Bains
  - Toulouse University Hospital, Toulouse
  - Clinique Teissier, Valenciennes
- Spain (6):
  - Hospital Vithas Xanit Internacional, Benalmádena, AN
  - Hospital Recoletas Campo Grande, Valladolid, CL
  - Consulta Respira, Mataró, CT
  - Hospital HM Montepríncipe, Boadilla del Monte, MD
  - Hospital HM Sanchinarro, Madrid, MD
  - Hospital HM Puerta del Sur, Móstoles, MD

IPD SHARING:
Plan to Share IPD: No